CLINICAL TRIAL: NCT00521950
Title: Pharmacogenetic Testing in the Clinical Setting: is Screening for TPMT Genotype a Cost-effective Treatment Strategy? - The First Prospective Randomized Controlled Trial Within the Dutch Health Care System.
Brief Title: Cost-effectiveness of TPMT Pharmacogenetics
Acronym: TOPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Marieke Coenen, PhD, Radboud University Medical Center
Organization: Radboud University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 945-07-606; CMO 2006/129; ABR NL13171.091.06
Record Dates: First submitted 2007-08-27; First posted 2007-08-28 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-03

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis
Keywords: Pharmacogenetics; Cost Effectiveness; Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis; Randomized Controlled Trials
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — Azathioprine; Mercaptopurine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention, TPMT genotyping (Experimental): Pre-treatment TPMT genotyping to optimize initial thiopurine treatment dose. Intervention is based on the genotype.
  Interventions: Genetic: TPMT genotyping; Drug: azathioprine or 6-mercaptopurine
- control (Active Comparator): Standard thiopurine treatment
  Interventions: Drug: azathioprine (AZA) or 6-mercaptopurine (6-MP)

INTERVENTIONS:
Genetic: TPMT genotyping; Drug: azathioprine or 6-mercaptopurine — Assessment of the polymorphisms G238C, G460A, and A719G in a venous blood sample to identify functional genetic variants (TPMT*2, *3A, *3C) of the TPMT gene (chromosome 6) associated with reduced or negligible TPMT enzyme activity.
  Patients are advised an initial treatment dose based on the enzyme activity:
  * Normal: AZA 2-2.5 mg/kg/day or 6-MP 1-1.5 mg/kg/day (standard care);
  * Reduced: AZA 1-1.25 mg/kg/day or 6-MP 0.5-0.75 mg/kg/day;
  * Negligible: AZA 0-0.2 mg/kg/day or 6-MP 0-0.1 mg/kg/day;
  Other Names: Imuran; Puri-Nethol
  Arms: Intervention, TPMT genotyping
Drug: azathioprine (AZA) or 6-mercaptopurine (6-MP) — Patients will be advised a standard initial treatment dose:
  * AZA 2-2.5 mg/kg/day or 6-MP 1-1.5 mg/kg/day (standard care);
  Other Names: Imuran; Puri-Nethol
  Arms: control

SUMMARY:
The purpose of this study is to determine whether thiopurine S-methyltransferase (TPMT) genotyping prior to thiopurine use is cost-effective in patients with inflammatory bowel disease (IBD) in need of immune suppression.

The study is designed to test the hypothesis that optimization of initial thiopurine dose based on pre-treatment TPMT genotyping will maximize treatment efficacy and minimize adverse drug reactions (ADRs) resulting in reduced costs.

DETAILED DESCRIPTION:
Immunosuppressives, e.g. azathioprine (AZA) and 6-mercaptopurine (6-MP), are important in induction of remission and long term treatment of (ulcerative) colitis and Crohn's disease when treatment with 5-aminosalicylates and corticosteroids fails. ADRs to immunosuppressive treatment, including myelosuppression and hepatotoxicity, are frequently (15-30%) observed. Genetic variation in the TPMT gene results in 10-11% of the general population in reduced and in 0.3-0.6% to negligible TPMT enzyme activity. In IBD patients, this genetic variation predicts 25-40% of the haematological ADRs necessitating tempering of thiopurine dose or discontinuation of treatment.

Pharmacogenetics aims at providing optimized drug treatment to patients by maximizing efficacy and minimizing adverse drug reactions (ADRs) based on genetic testing. Despite the proven value of pharmacogenetics in clinical practice, its use in medical care is still limited.

The best-established example of a pharmacogenetic test is genotyping of thiopurine S-methyltransferase (TPMT) in the treatment of patients with immunosuppressive thiopurines. Nonetheless, it is not used on a large scale in clinical practice so far, which might be due to: insufficient information transfer from research to clinic; lack of cost-effectiveness analyses (CEAs); lack of availability of (or access to) fast and/or cheap genotyping; or lack of test reimbursement by health insurance.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Diagnosis of a form of IBD
* Indication for azathioprine/6-MP treatment
* Patient giving (written) informed consent

Exclusion Criteria:

* Previous treatment with azathioprine/6-MP
* Co-prescription of allopurinol (this treatment blocks xanthine oxidase, an enzyme important for thiopurine metabolism)
* Baseline leukocyte count less then 3x10^9 per litre
* Reduced liver function at baseline
* Reduced renal function at baseline
* Known TPMT phenotype (enzyme activity / Therapeutic Drug Monitoring) or genotype
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 853 (Actual)
Dates: Start 2007-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Haematological adverse drug reactions | 0-5 months

SECONDARY OUTCOMES:
Non-haematological Adverse Drug Reactions | 0- 5 months
Clinical outcome (disease activity) | 5 months
Treatment compliance | 0 to 5 months
TPMT enzym activity | at baseline
Therapeutic Drug Monitoring of TPMT Metabolites | week 1 and 8
Health related quality of life | 5 months
Cost-efficacy | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Franke, PhD, Study Director — Radboud University Medical Center; Hans Scheffer, PhD, Study Chair — Radboud University Medical Center; Corine J van Marrewijk, MSc, Principal Investigator — Radboud University Medical Center; Dirk J de Jong, MD PhD, Principal Investigator — Radboud University Medical Center; Marieke JH Coenen, PhD, Study Chair — Radboud University Medical Center; Henk-Jan Guchelaar, PhD, Study Chair — Leiden UMC; Luc Derijks, PhD, Study Chair — Maxima MC Veldhoven; Olaf Klungel, PhD, Study Chair — UMC Utrecht; André Verbeek, PhD, Study Chair — Radboud University Medical Center; Sita Vermeulen, MSc, Study Chair — Radboud University Medical Center
Locations (3):
- Netherlands (3):
  - Radboud University Medical Center, Nijmegen, Gelderland
  - Bernhoven Hospital, Oss
  - Bernhoven Hospital, Veghel

REFERENCES:
- [Derived] Wong DR, Coenen MJ, Derijks LJ, Vermeulen SH, van Marrewijk CJ, Klungel OH, Scheffer H, Franke B, Guchelaar HJ, de Jong DJ, Engels LG, Verbeek AL, Hooymans PM; TOPIC Recruitment Team. Early prediction of thiopurine-induced hepatotoxicity in inflammatory bowel disease. Aliment Pharmacol Ther. 2017 Feb;45(3):391-402. doi: 10.1111/apt.13879. Epub 2016 Dec 12. PMID 27943397
- [Derived] Wong DR, Coenen MJ, Vermeulen SH, Derijks LJ, van Marrewijk CJ, Klungel OH, Scheffer H, Franke B, Guchelaar HJ, de Jong DJ, Engels LG, Verbeek AL, Hooymans PM; TOPIC recruitment team. Early Assessment of Thiopurine Metabolites Identifies Patients at Risk of Thiopurine-induced Leukopenia in Inflammatory Bowel Disease. J Crohns Colitis. 2017 Feb;11(2):175-184. doi: 10.1093/ecco-jcc/jjw130. Epub 2016 Jul 9. PMID 27402913
- [Derived] Coenen MJ, de Jong DJ, van Marrewijk CJ, Derijks LJ, Vermeulen SH, Wong DR, Klungel OH, Verbeek AL, Hooymans PM, Peters WH, te Morsche RH, Newman WG, Scheffer H, Guchelaar HJ, Franke B; TOPIC Recruitment Team. Identification of Patients With Variants in TPMT and Dose Reduction Reduces Hematologic Events During Thiopurine Treatment of Inflammatory Bowel Disease. Gastroenterology. 2015 Oct;149(4):907-17.e7. doi: 10.1053/j.gastro.2015.06.002. Epub 2015 Jun 11. PMID 26072396